CLINICAL TRIAL: NCT01903291
Title: A Multicenter, Open-Label, 12-Month Observational Study Evaluating the Clinical Effectiveness and Impact on Patient-Reported Outcomes of Oral Tecfidera™ (Dimethyl Fumarate) Delayed-Release Capsules in Patients With Relapsing Forms of Multiple Sclerosis After Suboptimal Response to Glatiramer Acetate
Brief Title: Effectiveness of DMF and Its Impact on PROs in Suboptimal GA Responders With RMS
Acronym: RESPOND
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 109MS404
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Relapsing Forms of Multiple Sclerosis
MeSH Terms: interventions — Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- dimethyl fumarate: To be taken according to the United States Prescribing Information (USPI)
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — As described in the treatment arm
  Other Names: Tecfidera; BG00012; DMF

SUMMARY:
The primary objective of the study is to estimate the annualized relapse rate (ARR) over a 12-month period in patients with relapsing forms of multiple sclerosis (MS) who are treated with dimethyl fumarate (DMF) after suboptimal response to glatiramer acetate (GA). The secondary objectives of this study in this study population are to assess the impact of DMF over a 12-month period on patient-reported outcomes (PROs) and health economic-related outcomes and to evaluate additional clinical outcomes at Month 12.

ELIGIBILITY:
Key Inclusion Criteria:

* Have the ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use Protected Health Information in accordance with national and local patient privacy regulations.
* Have the ability to read and understand written English.
* Have access to the internet and are able to complete online assessments on a computer
* Have a relapsing form of Multiple Sclerosis and satisfy the approved therapeutic indication for dimethyl fumarate (DMF) per the United States Prescribing Information (USPI).
* Are being treated for relapsing forms of multiple sclerosis (MS) with glatiramer acetate (GA) but, per the Prescribing Physician, have a suboptimal response (e.g., suboptimal efficacy, intolerance, or poor adherence) to GA or have stopped treatment with GA for relapsing forms of MS as a result of suboptimal response within 30 days of enrollment.
* Have decided to initiate treatment with dimethyl fumarate (DMF) under routine clinical care. The decision to initiate treatment with DMF must precede enrollment.
* Have a complete blood count (CBC) available within 6 months of initiation of treatment with dimethyl fumarate (DMF).

Key Exclusion Criteria:

* Are unwilling or unable to comply with study requirements, or, are deemed unsuitable for study participation at the discretion of the Prescribing Physician.
* Have major comorbid conditions that would preclude their participation in the study as determined by the Prescribing Physician.
* Have a history of malignancy. (Patients with basal cell carcinoma that has been completely excised prior to study entry remain eligible.)
* Have a history of and/or current serious infections.
* Are pregnant or breastfeeding, or are planning to become pregnant or breastfeed.
* Are receiving concomitant disease modifying therapies other than glatiramer acetate (GA) or have initiated treatment with a new disease-modifying therapy since discontinuation of glatiramer acetate (GA).
* Are currently enrolled in any other clinical studies, with the exception of the dimethyl fumarate (DMF) Pregnancy Registry.
* Have received prior treatment with dimethyl fumarate (DMF).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in male and female patients with relapsing forms of MS who satisfy the therapeutic indication for dimethyl fumarate (DMF) per the United States Prescribing Information, and who are suboptimal responders to glatiramer acetate (GA), as determined by the Prescribing Physician.
Sampling Method: Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2013-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Annualized Relapse Rate | 12 months

SECONDARY OUTCOMES:
Change in 14-item Treatment Satisfaction Questionnaire for Medication (TSQM-14) scores. | Baseline to 12 months
  TSQM-14 is an instrument to assess patient's satisfaction with medication, providing scores on four scales: Side effects, effectiveness, convenience and global satisfaction.
Change in Short-Form 36 (SF-36) scores. | Baseline to 12 months
  SF-36 is a self-administered, generic health status questionnaire consisting of 36 questions that measure 8 health concepts: physical functioning, role limitations due to physical problems, bodily pain, general health perception, vitality, social functioning, role limitations due to emotional problems and mental health.
Change in Modified Fatigue Impact Scale (MFIS-5) scores. | Baseline to 12 months
  MFIS-5 is a modified form of the Fatigue Impact Scale that consists of five questions that assess the impact of fatigue on physical, cognitive, and psychosocial functioning, with five response levels ranging from 0 ("Never") to 4 ("Almost always"). Total scores range from 0 to 20, with higher scores representing a greater impact of fatigue.
Change in Beck Depression Inventory (BDI-7) scores. | Baseline to 12 months
  BDI-7 is a self-report inventory for measuring the severity of depression on a 7-item scale.
Change in Work Productivity and Impairment Questionnaire: Multiple Sclerosis (WPAI-MS) scores. | Baseline to 12 months
  The Work Productivity and Activity Impairment (WPAI) questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteesism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Change in Morisky 8-item Medication Adherence Scale (MMAS-8) scores. | Baseline to 12 months
  MMAS-8 is a self-reporting tool to facilitate the identification of barriers to and behaviors associated with adherence to chronic medications. Scores on the MMAS-8 range from 0-8, with scores of less than 6 reflecting low adherence.
Change in Patient-reported Expanded Disability Status Scale (patient-reported EDSS) scores. | Baseline to 12 months
  The patient-reported EDSS measures disability status based on patient report of degree of difficulty in eight different functional areas (on a 4-point scale), and overall function, taking into account the eight areas and descriptions of gait.
Proportion of patients experiencing a relapse. | Baseline to 12 months
Proportion of patients with relapses associated with hospitalizations. | Baseline to 12 months
Proportion of patients with relapses associated with steroid use. | Baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (60):
- United States (60):
  - Research Site, Birmingham, Alabama
  - Research Site, Tuscon, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, San Jose, California
  - Research Site, Englewood, Colorado
  - Research Site, Dover, Delaware
  - Research Site, Jacksonville, Florida
  - Research Site, Lighthouse PT, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Franklin, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Lenexa, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Lexington, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Clinton Township, Michigan
  - Research Site, Muskegon, Michigan
  - Research Site, Golden Valley, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, Great Falls, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Freehold, New Jersey
  - Research Site, New York, New York
  - Research Site, Patchogue, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Centerville, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Greensburg, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Knoxville, Tennessee
  - Research Site, Round Rock, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Bellingham, Washington
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Neenah, Wisconsin

REFERENCES:
- [Derived] Repovic P, Robertson D, Kresa-Reahl K, Cohan SL, Su R, Avila R, Koulinska I, Mendoza JP. Effectiveness of Dimethyl Fumarate in Patients With Relapsing Multiple Sclerosis Switching After Suboptimal Response to Glatiramer Acetate, Including Patients With Early Multiple Sclerosis: Subgroup Analysis of RESPOND. Neurol Ther. 2021 Jun;10(1):169-182. doi: 10.1007/s40120-020-00223-2. Epub 2020 Nov 23. PMID 33225410
- [Derived] Kresa-Reahl K, Repovic P, Robertson D, Okwuokenye M, Meltzer L, Mendoza JP. Effectiveness of Delayed-release Dimethyl Fumarate on Clinical and Patient-reported Outcomes in Patients With Relapsing Multiple Sclerosis Switching From Glatiramer Acetate: RESPOND, a Prospective Observational Study. Clin Ther. 2018 Dec;40(12):2077-2087. doi: 10.1016/j.clinthera.2018.10.011. Epub 2018 Nov 22. PMID 30470580